CLINICAL TRIAL: NCT03128645
Title: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Brief Title: The Effect of the Abdominal Corset on Colonoscopy
Status: Completed | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ebubekir Gündeş, Gastroenterological Surgery, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2017/3/19
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Colonoscopy; Complete Colonoscopy; Cecum Intubation Time; İleum Intubation Time

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Standard method group
  Interventions: Device: Abdominal Corset
- Group 2: Abdominal corset group
  Interventions: Device: Abdominal Corset

INTERVENTIONS:
Device: Abdominal Corset — The patient's colonoscopy procedure in group 2 after randomization will be performed with the abdominal corset.

SUMMARY:
In patients with central obesity, the effect of the abdominal corset on colonoscopy completeness, cecum and ileum intubation time will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years, Meeting the central obesity criteria Cases where colonoscopy is performed under elective conditions

Exclusion Criteria:

* In case of emergency, The process is terminated due to bad bowel preparation, Inflammatory bowel disease, Serious arrhythmia, Chronic obstructive pulmonary disease Coronary artery disease The previous abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were remotely applying to our clinic and planned for colonoscopy according to ASGE colonoscopy indications.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Central Obesity | 01/04/2017- 01/06/2017
  BMI ≥ 30 (kg / m2), waist circumference> 102 cm in men and waist circumference> 88 cm in women
Cecum intubation time | 01/04/2017- 01/06/2017
  Insertion time of the colonoscope from anus to the cecum (second)
İleum intubation time | 01/04/2017- 01/06/2017
  Insertion time of the colonoscope from cecum to the ileum (second)

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Kosuyolu Yuksek Ihtisas Education and Research, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gundes E, Ofkeli O, Uzun O, Senger AS, Polat E, Duman M. Effect of Abdominal Corset on Completion of Colonoscopy and Cecal and Ileocecal Intubation Time in Patients with Central Obesity: A Prospective Randomized Controlled Trial. Ann Ital Chir. 2024;95(4):603-608. doi: 10.62713/aic.3348. PMID 39186356